CLINICAL TRIAL: NCT01941069
Title: Targeting School Climate and Children's Behavioral Health in Urban Schools
Brief Title: School Climate and Children's Behavioral Health
Acronym: Project Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Devereux Foundation, Pennsylvania (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The School District of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-009477; 5R01HD073430-02 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Consultation (LLS); Consultation and Coaching (HLS)
MeSH Terms: interventions — 6-chloro-2-(1-piperazinyl)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internalizing Disorders (Active Comparator): Students identified as being at-risk for or meeting criteria for Internalizing Disorders will assigned to this intervention arm. They will receive the FRIENDS for Life intervention. FRIENDS is a group Cognitive Behavioral Therapy (CBT) intervention, based on a theoretical model, which addresses cognitive, physiological and behavioral processes that are seen to interact in the development and perpetuation of excessive anxiety.
  Interventions: Behavioral: Friends for Life
- Externalizing Disorders (Active Comparator): Students identified as being at-risk for or meeting criteria for Externalizing Disorders will be assigned to this intervention arm. They will receive the Coping Power Program (CPP) intervention. CPP is a cognitive-behavioral, multi-component group intervention for elementary and middle school students at risk for externalizing behavior disorders. In addition to anger management, the CPP includes units on goal setting, emotional awareness, relaxation training, social skills training, problem solving, and handling peer pressure.
  Interventions: Behavioral: Coping Power Program

INTERVENTIONS:
Behavioral: Friends for Life — Friends for Life is a group CBT intervention, based on a theoretical model, which addresses cognitive, physiological and behavioral processes that are seen to interact in the development and perpetuation of excessive anxiety.
  Other Names: FRIENDS
  Arms: Internalizing Disorders
Behavioral: Coping Power Program — The Coping Power Program CPP is a cognitive-behavioral, multi-component group intervention for elementary and middle school students at risk for externalizing behavior disorders. In addition to anger management, the CPP includes units on goal setting, emotional awareness, relaxation training, social skills training, problem solving, and handling peer pressure.
  Other Names: CPP
  Arms: Externalizing Disorders

SUMMARY:
The overall purpose of this project is to determine whether school personnel implementing a two-tier School-wide Positive Behavior Support (SWPBS, an evidence based intervention) program for typically developing children as well as children with, or at risk for, externalizing or anxiety disorders can implement the components of the program with the same level of fidelity, integrity and clinical effectiveness when they receive a low level of support (consultation) from their coaches and supervisors as they can with a high level of support (consultation and coaching).

DETAILED DESCRIPTION:
Demonstrating that school personnel can implement evidence based interventions (EBIs) for externalizing and anxiety problems with a high degree of fidelity, integrity and clinical effectiveness could spur more initiatives toward the adoption of EBIs in urban schools, thus further lowering health disparities in these settings. The overall purpose of this project is to determine whether school personnel implementing a two-tier School-wide Positive Behavior Support (SWPBS, an evidence based intervention) program for typically developing children as well as children with, or at risk for, externalizing or anxiety disorders can implement the components of the program with the same level of fidelity, integrity and clinical effectiveness when they receive a low level of support (consultation) from their coaches and supervisors as they can with a high level of support (consultation and coaching). This study will target six schools within the Philadelphia School District (PSD). Within those 6 schools, research participants will consist of students (grades 4-8) and school staff members. The investigators will evaluate 1) the effectiveness of SWPBS with consultation and coaching, as compared to the baseline and to SWPBS with consultation only; in reducing office discipline referrals (ODRs) and improving school climate, and children's grades, diagnostic status, symptom severity and impairment; 2) the effectiveness of the SWPBS with consultation and coaching, as compared to SWPBS with consultation only, in increasing program fidelity and integrity.

ELIGIBILITY:
Inclusion Criteria:

* All 6 participating schools are included in Tier 1.
* The inclusion criteria for Tier 2 includes children in grades 3-8, who are referred by a school staff member because of behavioral or emotional difficulties or because they have received 3 or more Office Discipline Referrals. Children who consent to participate in the project.

Exclusion Criteria:

* There are no exclusion criteria for Tier 1.
* The exclusion criteria for Tier 2 include any child in grades 3-8 whose family chooses not to consent to screening or participate in the intervention, has Special Education classification of "Intellectual Disability", who is not able to communicate in English, or has a history of psychotic or autistic spectrum disorders.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 437 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Level of Support During Implementation | 48 months
  To determine whether program fidelity and integrity for Tier 1 (for all students) and Tier 2 (for at risk and high risk students) would differ between schools receiving a high level of support (consultation and coaching) and schools receiving a low level of support (consultation) for program implementers.

SECONDARY OUTCOMES:
Cost Benefit Analyses | 48 months
  The secondary objectives are to determine the incremental cost-effectiveness of SWPBS HLS (consultation and coaching) versus SWPBS LLS (consultation).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo B. Eiraldi, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The School District of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Eiraldi R, Mautone JA, Khanna MS, Power TJ, Orapallo A, Cacia J, Schwartz BS, McCurdy B, Keiffer J, Paidipati C, Kanine R, Abraham M, Tulio S, Swift L, Bressler SN, Cabello B, Jawad AF. Group CBT for Externalizing Disorders in Urban Schools: Effect of Training Strategy on Treatment Fidelity and Child Outcomes. Behav Ther. 2018 Jul;49(4):538-550. doi: 10.1016/j.beth.2018.01.001. Epub 2018 Jan 6. PMID 29937256
- [Derived] Eiraldi R, McCurdy B, Khanna M, Mautone J, Jawad AF, Power T, Cidav Z, Cacia J, Sugai G. A cluster randomized trial to evaluate external support for the implementation of positive behavioral interventions and supports by school personnel. Implement Sci. 2014 Jan 15;9:12. doi: 10.1186/1748-5908-9-12. PMID 24428904